CLINICAL TRIAL: NCT03096886
Title: Novel Neural Circuit Biomarkers of Major Depression Response to Computer-augmented CBT
Brief Title: Novel Neural Circuit Biomarkers of Major Depression Response to CCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH110939-01A1 (NIH)
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Depression; Major Depressive Disorder; Depressive Disorder; Depression, Unipolar
Keywords: Cognitive Behavioral Therapy; Computer-Assisted Cognitive Behavioral Therapy; Computer-Augmented Cognitive Behavioral Therapy; CBT; Computer-Assisted CBT; Computer-Augmented CBT
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: This is a 3-arm, parallel study design. Individuals presenting with MDD will be randomized into either Arm 1: 8 weeks of Computer-Augmented Cognitive Behavioral Therapy (CCBT) Immediately or Arm 2: Waitlist up to 4 weeks followed by 8 weeks of CCBT. Arm 3 is a no treatment arm for matched comparison participants (i.e., healthy controls).
Who Masked: Outcomes Assessor
Masking Description: An experienced clinical evaluator with established reliability will assess patients pre-treatment and biweekly during CCBT treatment (Weeks 1, 2, 4, 6, 8, 9 of CCBT). All evaluations will be conducted without knowledge of treatment assignment. The evaluator will assess symptom severity according to the MADRS and Hamilton Rating Scale for Depression (HAM-D). Evaluators will have offices remote to the day-to-day operations of the treatment study and will not participate in weekly study management meetings in order to help preserve the blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early CCBT (Experimental): Intervention: Computer-Augmented Cognitive Behavioral Therapy
  Half of participants presenting with MDD will be randomized to receive 8 weeks of Computer-Augmented Cognitive Behavior Therapy (CCBT) immediately after completing pre-treatment assessments; imaging data will be collected pre- and post-treatment.
  Interventions: Behavioral: Computer-Augmented Cognitive Behavioral Therapy
- Late CCBT (Experimental): Intervention: Waitlist followed by Computer-Augmented Cognitive Behavioral Therapy
  Half of participants presenting with MDD will be randomized to be waitlisted for up to 4 weeks and will receive CCBT within 4 weeks; imaging data will also be collected pre--treatment, following waitlist, and post-treatment of CCBT.
  This arm will serve as the equivalent of a "placebo comparator" arm during the waitlist; and then as an experimental arm when receiving 8 weeks of CCBT treatment.
  Interventions: Behavioral: Computer-Augmented Cognitive Behavioral Therapy
- Matched Comparison (No Intervention): No Intervention: Matched Comparison
  Healthy controls will act as a matched comparator. Participants will complete pre-treatment assessments and imaging.

INTERVENTIONS:
Behavioral: Computer-Augmented Cognitive Behavioral Therapy — The model of CCBT, "Good Days Ahead" (GDA) will be utilized, it has been found that it is not inferior to CBT in MDD treatment efficacy. CCBT participants will complete 9 modules of the GDA program, including 240 minutes of computer training; participants will also meet with a therapist on 6 occasions for a total of 180 minutes of clinician administered cognitive behavioral therapy.
  Other Names: CCBT; Computer-Assisted Cognitive Behavioral Therapy
  Arms: Early CCBT; Late CCBT

SUMMARY:
The purpose of the study is to learn more about computer-assisted cognitive behavioral therapy or "CCBT" and to examine connections in the brains of patients with depression. CCBT is approved by the FDA as a form of treatment for depression. It is done partly on the computer and partly with a therapist.

This study will enroll participants with depression and participants without depression. The investigators will recruit a total of 100 participants: 80 with Major Depressive Disorder (MDD) and 50 matched comparison participants.

Healthy control subjects will participate for approximately 8 weeks.

All MDD participants will receive CCBT. Half of the MDD participants will all receive computer-augmented skills training with the Good Days Ahead (GDA) protocol immediately (Early CCBT). Early CCBT subjects will participate for approximately 8 weeks. The other half of the MDD participants initially will be randomized to a waitlist of up to 4 weeks and subsequently will receive CCBT treatment (Late CCBT). Late CCBT subjects will participate for approximately 12 weeks.

All participants are asked to complete a screening, which includes a series of clinical interviews and self-report questionnaires about the individual's thoughts, moods, and behaviors. All participants are asked to wear an actigraph, which is a watch-like device that measures activity levels. Additionally, participants are asked to completed short questions and have their activity levels monitored through phone app(s).

All participants (Healthy Control and MDD participants) will receive functional magnetic resonance imaging (fMRI) scanning at baseline. Early CCBT participants will receive fMRI scanning after 8 weeks of CCBT, and Late CCBT participants will receive fMRI scanning at the conclusion of the waitlist and after the 8-week course of CCBT. Brain activity will be compared between MDD and controls at baseline and between Early CCBT vs Late CCBT. The 2nd and 3rd brain scans of Late CCBT participants at the end of the waitlist and 8-week course of CCBT, respectively, will allow within-subject comparison of CCBT vs Waitlist treatment effects.

This clinical trial has two IRB protocol numbers: 826910 and 832295. The data collected through both protocol numbers will be analyzed together to accomplish the target of 100 subjects for this clinical trial.

DETAILED DESCRIPTION:
This study is a randomized study. 80 subjects with MDD will be randomly assigned (1:1) to immediately receive 8 weeks of CCBT or delayed treatment, consisting of up to 4 weeks of waitlist, followed by 8 weeks of CCBT. 50 healthy controls of similar age/sex will be recruited to serve as a comparison group for baseline magnetic resonance imaging (MRI) scanning.

The study will enroll subjects for approximately 4 years (~2 subjects per month for 48 months). The length of subject participation will vary based on what group the participants are randomized to. Healthy controls will participate for approximately 8 weeks. Subjects with MDD who were randomized to Early CCBT will participate for approximately 8 weeks; subjects with MDD who were randomized to Late CCBT will participate for approximately 12 weeks. Variability in the study duration for each group depends on each subjects' personal availability for visits and the availability of the magnetic resonance scanner.

Potential participants will complete a phone screen to determine eligibility. If the individual is eligible, the individual will be scheduled for an in-person screening visit. Information collected during the phone screening will not be used in the data analysis; phone screening information will be collected and retained in REDCap. Remote contact options are available as needed/possible.

Screening Visit - all participants will have the study described to them in detail, including the risks and study procedures as outlined in the informed consent form and will sign the informed consent form (ICF) and HIPAA authorization, prior to any study procedures being completed. Participants will be screened for symptoms of psychological disorders and severity of major depressive symptoms by a trained research team member.

If determined eligible, HEALTHY CONTROLS will be scheduled for return to complete an fMRI scan and baseline visit, in which self-report measures, including reports of mood, behavior, and thoughts will be collected, as well as neuropsychological testing. The HIPAA-compliant phone app Beiwe and actigraph setup will take place during the baseline visit. Participants will complete mood monitoring questions on the phone app and also have their activity levels monitored by the phone app and the actigraph for the duration of the study.

If determined eligible at screening, MDD (EXPERIMENTAL GROUP) participants will be randomized (1:1) as follows: One half of the depressed participants will be randomized to receive 8 weeks of CCBT immediately after completing pretreatment assessments and the remainder will be randomized to a waitlist of up to 4 weeks followed by 8 weeks of CCBT.

MDD, EARLY CCBT GROUP Early CCBT participants will be scheduled for return to complete an fMRI scan at the baseline visit, in which self-report measures, including reports of mood, behavior, and thoughts will be collected, as well as neuropsychological testing. The phone apps Beiwe and Ethica and actigraph setup will take place during the baseline visit. Participants will complete mood monitoring questions on the phone apps and also have their activity levels monitored by the phone app and the actigraph for the duration of the study. Participants will complete Good Days Ahead (GDA) computer training throughout the 8 weeks of CCBT, and having 6 encounters with a licensed psychologist/psychiatrist. Additionally, outcome measures will be assessed by an independent clinical evaluator (without knowledge of treatment assignment) every other week. As soon as can be arranged after Week 9 of CCBT treatment (last CCBT Clinical Contact), participants will return to complete an fMRI scan and end of study visit, in which self-report measures, including reports of mood, behavior, and thoughts will be collected, as well as neuropsychological testing.

MDD, LATE CCBT GROUP Late CCBT participants will be scheduled for return to complete an fMRI scan and baseline visit, in which self-report measures, including reports of mood, behavior, and thoughts will be collected, as well as neuropsychological testing. The phone apps Beiwe and Ethica and actigraph setup will take place during the baseline visit. During the 2-4 week waitlist phase, participants will complete mood monitoring questions on the phone apps and also have their activity levels monitored by the phone app and the actigraph.

At the conclusion of the waitlist of up to 4 weeks, participants will complete a second fMRI scan and complete self-report measures, including reports of mood, behavior, and thoughts will be collected, as well as neuropsychological testing.

Participants will then enter the CCBT phase and will complete Good Days Ahead (GDA) computer training throughout the 8 weeks of CCBT. They will have 6 encounters with a licensed psychologist/psychiatrist at multiple time points during this period. Additionally, outcome measures will be assessed by an independent clinical evaluator (without knowledge of treatment assignment) every other week during this study phase. At Week 9 of CCBT treatment (last CCBT Clinical Contact), participants will complete a 1-hour fMRI scan and self-report measures, including reports of mood, behavior, and thoughts will be collected, as well as neuropsychological testing.

This clinical trial has two IRB protocol numbers: 826910 and 832295. The data collected through both protocol numbers will be analyzed together to accomplish the target of 130 subjects for this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 - 60 years old, gender inclusive
2. Willing to not take psychotropic medications for the duration of the study
3. Fluent in English (both verbally and written)
4. Able and willing to provide consent
5. Has reliable access to a private computer or electronic tablet
6. Owns a smart phone (iPhone or Android) with ability to download apps

Experimental group 1) Diagnosis of MDD, experiencing current episode as determined by SCID-5 2) Current major depressive episode of moderate severity, as determined by MADRS score of 20 or higher

Control group 1) No history of MDD in lifetime 2) No indication of current, significant depressive symptoms, as determined by MADRS score of 8 or lower

Exclusion Criteria:

1. Diagnosis of severe or poorly controlled concurrent medical disorders that may cause depression or require medication that could cause depressive symptoms
2. Unwilling to provide informed consent
3. Diagnosis of concurrent DSM-5 (SCID) psychiatric disorders: any psychotic or organic mental disorder, bipolar disorder, active alcohol or drug dependence, primary anxiety disorder or primary eating disorders (primary refers to the diagnosis associated with the most functional impairment)
4. Diagnosed (DSM-5 criteria) by the clinical coordinator with attention deficit hyperactivity disorder, learning disorder, borderline personality disorder, antisocial personality disorder, or paranoid personality disorder
5. Cannot complete questionnaires written in English
6. Have not completed at least a 10th grade education or a general education degree (GED)
7. Represent an active suicide risk
8. Centrally acting antiadrenergic agents
9. Have MRI contraindications (e.g., foreign metallic implants, pacemaker, severe claustrophobia)
10. Currently demonstrating a response to antidepressant/psychotropic medication (besides SSRIs, which are acceptable if use has been stable over at least a 2 month period)

Experimental group 1) Score less than 20 on the MADRS at either initial interview or 18 at second interview 2) Have previously failed to respond to a trial of at least 8 weeks of CBT conducted by a certified therapist) 3) Are currently demonstration a response to antidepressant/psychotropic medication besides SSRIs, which are acceptable if use has been stable over at least a 2 month period (individuals taking a psychotropic medication may stop taking it for the purpose of the study ONLY if they are not receiving clinical benefits from taking it and after meeting with one of the study doctors to discuss the risks/benefits of discontinuing the medication and other treatment options)

Control group 1) Must have no lifetime history of a major depressive episode 2) Must score below 8 on the MADRS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette I Sheline, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shou H, Yang Z, Satterthwaite TD, Cook PA, Bruce SE, Shinohara RT, Rosenberg B, Sheline YI. Cognitive behavioral therapy increases amygdala connectivity with the cognitive control network in both MDD and PTSD. Neuroimage Clin. 2017 Jan 27;14:464-470. doi: 10.1016/j.nicl.2017.01.030. eCollection 2017. PMID 28275546
- [Background] Newman MG, Szkodny LE, Llera SJ, Przeworski A. A review of technology-assisted self-help and minimal contact therapies for anxiety and depression: is human contact necessary for therapeutic efficacy? Clin Psychol Rev. 2011 Feb;31(1):89-103. doi: 10.1016/j.cpr.2010.09.008. Epub 2010 Oct 14. PMID 21130939
- [Background] Vittengl JR, Clark LA, Jarrett RB. Continuation-phase cognitive therapy's effects on remission and recovery from depression. J Consult Clin Psychol. 2009 Apr;77(2):367-71. doi: 10.1037/a0015238. PMID 19309197
- [Background] Biesheuvel-Leliefeld KE, Kok GD, Bockting CL, Cuijpers P, Hollon SD, van Marwijk HW, Smit F. Effectiveness of psychological interventions in preventing recurrence of depressive disorder: meta-analysis and meta-regression. J Affect Disord. 2015 Mar 15;174:400-10. doi: 10.1016/j.jad.2014.12.016. Epub 2014 Dec 13. PMID 25553400
- [Background] Seligman ME. The effectiveness of psychotherapy. The Consumer Reports study. Am Psychol. 1995 Dec;50(12):965-74. doi: 10.1037//0003-066x.50.12.965. PMID 8561380
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Wright JH, Wright AS, Albano AM, Basco MR, Goldsmith LJ, Raffield T, Otto MW. Computer-assisted cognitive therapy for depression: maintaining efficacy while reducing therapist time. Am J Psychiatry. 2005 Jun;162(6):1158-64. doi: 10.1176/appi.ajp.162.6.1158. PMID 15930065
- [Background] Eells TD, Barrett MS, Wright JH, Thase M. Computer-assisted cognitive-behavior therapy for depression. Psychotherapy (Chic). 2014 Jun;51(2):191-7. doi: 10.1037/a0032406. Epub 2013 Sep 23. PMID 24059735
- [Background] Korgaonkar MS, Fornito A, Williams LM, Grieve SM. Abnormal structural networks characterize major depressive disorder: a connectome analysis. Biol Psychiatry. 2014 Oct 1;76(7):567-74. doi: 10.1016/j.biopsych.2014.02.018. Epub 2014 Mar 6. PMID 24690111
- [Background] Mayberg HS. Limbic-cortical dysregulation: a proposed model of depression. J Neuropsychiatry Clin Neurosci. 1997 Summer;9(3):471-81. doi: 10.1176/jnp.9.3.471. PMID 9276848
- [Background] Drevets WC, Price JL, Furey ML. Brain structural and functional abnormalities in mood disorders: implications for neurocircuitry models of depression. Brain Struct Funct. 2008 Sep;213(1-2):93-118. doi: 10.1007/s00429-008-0189-x. Epub 2008 Aug 13. PMID 18704495
- [Background] Sheline YI, Barch DM, Donnelly JM, Ollinger JM, Snyder AZ, Mintun MA. Increased amygdala response to masked emotional faces in depressed subjects resolves with antidepressant treatment: an fMRI study. Biol Psychiatry. 2001 Nov 1;50(9):651-8. doi: 10.1016/s0006-3223(01)01263-x. PMID 11704071
- [Background] Hamilton JP, Etkin A, Furman DJ, Lemus MG, Johnson RF, Gotlib IH. Functional neuroimaging of major depressive disorder: a meta-analysis and new integration of base line activation and neural response data. Am J Psychiatry. 2012 Jul;169(7):693-703. doi: 10.1176/appi.ajp.2012.11071105. PMID 22535198
- [Background] Zhang J, Wang J, Wu Q, Kuang W, Huang X, He Y, Gong Q. Disrupted brain connectivity networks in drug-naive, first-episode major depressive disorder. Biol Psychiatry. 2011 Aug 15;70(4):334-42. doi: 10.1016/j.biopsych.2011.05.018. PMID 21791259
- [Background] Kaiser M. A tutorial in connectome analysis: topological and spatial features of brain networks. Neuroimage. 2011 Aug 1;57(3):892-907. doi: 10.1016/j.neuroimage.2011.05.025. Epub 2011 May 14. PMID 21605688
- [Background] Fales CL, Barch DM, Rundle MM, Mintun MA, Snyder AZ, Cohen JD, Mathews J, Sheline YI. Altered emotional interference processing in affective and cognitive-control brain circuitry in major depression. Biol Psychiatry. 2008 Feb 15;63(4):377-84. doi: 10.1016/j.biopsych.2007.06.012. Epub 2007 Aug 24. PMID 17719567
- [Background] Satterthwaite TD, Cook PA, Bruce SE, Conway C, Mikkelsen E, Satchell E, Vandekar SN, Durbin T, Shinohara RT, Sheline YI. Dimensional depression severity in women with major depression and post-traumatic stress disorder correlates with fronto-amygdalar hypoconnectivty. Mol Psychiatry. 2016 Jul;21(7):894-902. doi: 10.1038/mp.2015.149. Epub 2015 Sep 29. PMID 26416545
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788

RESULTS

PARTICIPANT FLOW:
Groups:
- Early CCBT: Intervention: Computer-Augmented Cognitive Behavioral Therapy
  Half of participants presenting with MDD will be randomized to receive 8 weeks of Computer-Augmented Cognitive Behavior Therapy (CCBT) immediately after completing pre-treatment assessments; imaging data will be collected pre- and post-treatment.
  Computer-Augmented Cognitive Behavioral Therapy: The model of CCBT, "Good Days Ahead" (GDA) will be utilized, it has been found that it is not inferior to CBT in MDD treatment efficacy. CCBT participants will complete 9 modules of the GDA program, including 240 minutes of computer training; participants will also meet with a therapist on 6 occasions for a total of 180 minutes of clinician administered cognitive behavioral therapy.
- Late CCBT: Intervention: Waitlist followed by Computer-Augmented Cognitive Behavioral Therapy
  Half of participants presenting with MDD will be randomized to be waitlisted for up to 4 weeks and will receive CCBT within 4 weeks; imaging data will also be collected pre--treatment, following waitlist, and post-treatment of CCBT.
  This arm will serve as the equivalent of a "placebo comparator" arm during the waitlist; and then as an experimental arm when receiving 8 weeks of CCBT treatment.
  Computer-Augmented Cognitive Behavioral Therapy: The model of CCBT, "Good Days Ahead" (GDA) will be utilized, it has been found that it is not inferior to CBT in MDD treatment efficacy. CCBT participants will complete 9 modules of the GDA program, including 240 minutes of computer training; participants will also meet with a therapist on 6 occasions for a total of 180 minutes of clinician administered cognitive behavioral therapy.
Period: Overall Study
Arm/Group | Early CCBT | Late CCBT | Matched Comparison
Started | 38 | 44 | 50
Completed | 30 | 30 | 40
Not Completed | 8 | 14 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early CCBT | Late CCBT | Matched Comparison | Total
Number analyzed (Participants) | 30 | 30 | 40 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 40 | 100
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (7.98) | 29.1 (9.5) | 27.7 (7.9) | 28.4 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 26 | 68
  Male | 9 | 9 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 10
  Not Hispanic or Latino | 26 | 26 | 38 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 5 | 3 | 9 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 8 | 23
  White | 16 | 18 | 22 | 56
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 40 | 100

OUTCOME MEASURES:

1. Primary Outcome: Resting State Functional Connectivity: MDD vs Controls
Description: Compare baseline resting state functional connectivity and task-induced activity between MDD (early and late CCBT combined) and controls. The connectivity values were Z-normalized Pearson's r values. Specifically, time series values were averaged across all voxels within each given Region Of Interest (ROI) (Left Dorsolateral Prefrontal Cortex and Subgenual Anterior Cingulate Cortex). For each study visit for each participant, the resulting region-wise time series values were then correlated with those from another ROI using a Pearson correlation. This correlation coefficient was then Z-normalized to yield the connectivity value. Improvement was defined as connectivity that is closer to negative (less positive). There is no relevant clinical threshold.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Z normalized correlation
Arm/Group | Early CCBT | Late CCBT | Matched Comparison
Number analyzed (Participants) | 36 | 36 | 40
Z normalized correlation | .51 (.21) | .65 (.21) | .54 (.17)

2. Secondary Outcome: Resting State Functional Connectivity: Immediate CCBT vs Waitlist Followed by CCBT
Description: Assess CCBT treatment effects on resting state functional connectivity and task-induced activity in MDD comparing Immediate CCBT treatment vs Waitlist followed by CCBT at 8 weeks. The connectivity values were Z-normalized Pearson's r values. Specifically, time series values were averaged across all voxels within each given Region Of Interest (ROI) (Left Dorsolateral Prefrontal Cortex and Subgenual Anterior Cingulate Cortex). For each study visit for each participant, the resulting region-wise time series values were then correlated with those from another ROI using a Pearson correlation. This correlation coefficient was then Z-normalized to yield the connectivity value. Improvement was defined as connectivity that is closer to negative (less positive). There is no relevant clinical threshold.
Time Frame: Week 8
Population: This data was only collected from the Early CCBT group and the Late CCBT group. It was not collected from the Matched Comparison group.
Measure: Mean (Standard Deviation); unit: Z normalized correlation
Arm/Group | Early CCBT | Late CCBT
Number analyzed (Participants) | 30 | 32
Z normalized correlation | .46 (.17) | .57 (.18)

ADVERSE EVENTS:
Time Frame: 3-6 months depending on how long and which group the participant was enrolled in.
Arm/Group | Early CCBT | Late CCBT | Matched Comparison
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/44 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/44 | 0/50
Other Adverse Events (participants affected / at risk) | 0/38 | 0/44 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03096886/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT03096886/ICF_001.pdf